CLINICAL TRIAL: NCT03978559
Title: A Prospective Randomized Controlled Study to Compare Efficacy of Caspofungin Combined With Trimethoprim-sulfamethoxazole Versus Trimethoprim/Sulfamethoxazole as First-line Therapy in Non-HIV Patients With Severe Pneumocystis Pneumonia
Brief Title: Trimethoprim/Sulfamethoxazole Combined With Caspofungin as First-line Therapy in PCP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bin Du (Other)
Responsible Party: Sponsor-Investigator, Bin Du, Director, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICU-PCP
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Pneumocystis Pneumonia
MeSH Terms: conditions — Pneumonia, Pneumocystis | interventions — Caspofungin; Sulfisoxazole; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAS with TMP/SMZ (Experimental)
  Interventions: Drug: caspofungin; Drug: TMP/SMZ(trimethoprim/sulfisoxazole); Drug: Methylprednisolone
- TMP/SMZ (Active Comparator)
  Interventions: Drug: TMP/SMZ(trimethoprim/sulfisoxazole); Drug: Methylprednisolone

INTERVENTIONS:
Drug: caspofungin — caspofungin 70mg ivdrip the first day, then 50mg ivdrip qd for 21days
  Arms: CAS with TMP/SMZ
Drug: TMP/SMZ(trimethoprim/sulfisoxazole) — TMP:15mg/kg/d for 21 days +SMZ:75mg/kg/d for 21days
Drug: Methylprednisolone — 40mg ivdrip q12h for 5 days , then 40mg ivdrip qd for 5 days , 20mg for 11 days

SUMMARY:
This is a prospective, randomized clinical trial. During the study, non-HIV patients who are admitted to ICU due to Pneumocystic pneumonia (PCP) and have not received anti-PCP therapy or have received therapy less than 48hrs will be randomized (1:1) to received caspofungin combined with trimethoprim-sulfamethoxazole or trimethoprim-sulfamethoxazole alone.

The aim of this study is to compare the effectiveness of caspofungin combined with trimethoprim-sulfamethoxazole with that of conventional therapy (trimethoprim-sulfamethoxazole alone) as first-line therapy in the treatment of severe Pneumocystis pneumonia (PCP) in non-HIV patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Non-HIV immunosuppressed patients admitted to the ICU
3. confirmed or suspect PCP

3) Not receiving anti-PCP treatment or anti-PCP treatment < 48 hours

Exclusion Criteria:

1. Age less than 18 years old
2. Known pregnancy
3. allergy to TMP/SMZ or caspofungin
4. Decision to withhold life-sustaining treatment
5. Patients with advanced pulmonary fibrosis
6. severe liver dysfunction(Child-Pugh C )

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-07-08 (Estimated)

PRIMARY OUTCOMES:
mortality to day 28 | 28 days after randomization
  The percentage of subjects death at study day 28. Those subjects discharged from ICU prior to day 28 were counted as alive at day 28

SECONDARY OUTCOMES:
ICU Free Days to day 28 | 28 days after randomization
  defined as the number of days between randomization and day 28 in which the patient is not in the ICU (for any part of a day)
Mean Ventilator Free Days to day 28 | 28 days after randomization
  Ventilator-free days is defined to be 28 days minus the duration of mechanical ventilation through day 28. Participants who do not survive to day 28 are assigned zero ventilator-free days.
ICU mortality | through ICU discharge, an average of 14 days
  The percentage of death subjects at ICU discharge
hospital mortality | through hospital discharge, an average of 28 days
  The percentage of death subjects at hospital discharge
PO2/FiO2 on day 7, 21 | day 7, 21 after randomization
  the change of PO2/FiO2 between baseline and day7, 21
serum (1,3)-β-D gluca level on day 3, 7, 21 | day3, 7, 21 after randomization
  the change of (1,3)-β-D glucan level between baseline and day3, 7, 21
PCP-DNA negative conversion rate in alveolar lavage fluid on day 7 after randomization | day 7 after randomization
  the percentage of PCP-DNA negative after 7days treatment
SOFA | day3, 7, 21 after randomization
  respiratory dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score for respiratory system
BALF cytokines level on day3, 7, 21 | day3, 7, 21 after randomization
  the change of cytokines in bronchoalveolar lavage fluid (BALF) level between baseline and day7, day21
adverse events | till 21 days after randomization
  incidence, duration and severity of adverse events
serious adverse events | till 21 days after randomization
  incidence, duration and severity of serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- MICU of Peking Union Medical College, Beijing, China